CLINICAL TRIAL: NCT01853683
Title: Interval Appendectomy in Children, is it Really Necessary? A Randomized, Noninferiority Trial
Brief Title: Is Interval Appendectomy Necessary?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Ahmed Nasr, Principal Investigator, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/02E
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Appendicitis
Keywords: General Surgery
MeSH Terms: conditions — Appendicitis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative Management (Experimental): Children randomized to conservative management will be seen in the clinic 6-10 weeks after discharge and phoned to follow up every 3 month for a total follow-up of a year. Family will be instructed to come back to the hospital or call the treating physician if the child develops any abdominal pain or fever.
  Interventions: Procedure: Conservative Management
- Operative Management (Active Comparator): Children randomized to IA will be scheduled for an interval appendectomy 6-10 weeks after discharge, and will be seen in the clinic 6-8 weeks following the interval appendectomy and phoned for follow-up every 3 month for a total of one year.
  Interventions: Procedure: Operative Management

INTERVENTIONS:
Procedure: Conservative Management
  Arms: Conservative Management
Procedure: Operative Management
  Arms: Operative Management

SUMMARY:
Appendicitis is one of the most common surgical problems in children, with 20-35% of patients having perforated by the time they present to a doctor. In these cases, the patient is often treated non-surgically with antibiotics. Once a patient has improved, it is not known whether it is better to perform an interval appendectomy (IA) or to continue a watchful waiting approach. The purpose of this trial is to determine if expectant nonoperative management (watchful waiting) is not inferior compared to IA management after successful conservative treatment of appendiceal mass at admission.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age
* Perforated appendicitis where the treating physician chooses to follow the conservative approach rather than performing an immediate appendectomy

Exclusion Criteria:

* Uncertainty about the diagnosis
* The need for laparotomy/laparoscopy for another reason
* Perforated appendicitis with diffuse abdominal fluid on imaging associated with a clinical picture of severe sepsis
* Another medical condition that may affect the decision to operate e.g., inflammatory bowel disease
* A comorbidity or chronic illness that contraindicates the watchful waiting approach, e.g, diabetes or cardiac problems

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recurrent appendicitis for the conservative group | During a year of follow-up
Operative complications for the operative group | During a year of follow-up

SECONDARY OUTCOMES:
Duration of hospital stay | This is the patients' original hospital stay, and re-admission for interval appendectomy when applicable, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nasr, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada